CLINICAL TRIAL: NCT03422133
Title: A Patient-oriented Risk Communication Tool to Improve Patient Experience, Knowledge and Outcomes After Elective Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20170737-01H
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Implementation Phase: Participants in this group (before the eHealth app is implemented in the PAU) will be English or French speaking patients, aged 18 and older, scheduled for major non-cardiac elective surgery.
  Patients will be recruited using standardized procedures, and process and outcome measures will be recorded using the same tools and methods in both study phases to decrease the risk of measurement and selection bias.
- Post-Implementation Phase: Participants in this group (after the eHealth app is implemented in the PAU) will be English or French speaking patients, aged 18 and older, scheduled for major non-cardiac elective surgery.
  Interventions: Other: Patient-oriented, personalized risk communication eHealth application

INTERVENTIONS:
Other: Patient-oriented, personalized risk communication eHealth application — The application features simple and consistent design, large well-lit buttons that tolerate tremor, and simple language. The process will be applied in preoperative clinics at The Ottawa Hospital (TOH), where patients will be asked to provide their personal health history through a series of questions already used on our TOH preoperative health screener. These values will then populate the NSQIP Universal Risk Calculator, which we have calibrated to TOH data, to generate personalized risks of mortality, serious complications, and hospital length of stay. These risk estimates will be communicated directly to the patient using absolute risk estimates represented pictorially (best practice for risk communication to patients). Risk estimates will also be provided to the patient's clinician.
  Groups: Post-Implementation Phase

SUMMARY:
Many people have inpatient surgery each day. Most people will have no complications but some will have minor or serious complications. The risk of having complications can vary from one person to another depending on personal factors such as; age, medical conditions such as diabetes and whether someone smokes or takes certain medications.

The Investigators have learned that people want more information about their surgeries, both the general information about the risk for complications, but also more specific information about whether they are personally more or less likely to have complications. Patients are also interested in practical information such as how long they might stay in the hospital and what the recovery period will be like for them. Receiving more information can help decrease a person's level of anxiety about their surgery.

The Investigators are doing this study with the assistance of the mHealth Lab at The Ottawa Hospital (a team that develops simple technologies for managing health information). The Investigators will implement and evaluate a novel, innovative tablet-based, patient-oriented risk communication application to evaluate patient knowledge of their own surgical risk before and after their visit to the Pre-Admission Unit (PAU). The Investigators will also be exploring any potential levels of anxiety before and after the PAU visit, in addition to patient satisfaction with their PAU visit.

The Investigators hypothesize that it will: improve patient knowledge and experience, not increase anxiety, be acceptable to patients and clinicians, and will improve care efficiency for TOH surgical patients.

DETAILED DESCRIPTION:
One and a half million Canadians have inpatient surgery every year, and many experience serious complications. Research shows that patient-specific risks are not routinely or effectively communicated to patients before surgery, despite the requirement for such information to be included as part of the informed consent process, and clear recommendations from best practice guidelines.

Mobile health technology can address this gap by engaging and empowering patients to provide their own health data to generate personalized risk estimates. Using a tablet-based platform, these risk estimates can then be communicated to patients in a format that is appealing and understandable. However, such an application and process do not exist.

The Investigators will address this knowledge gap through the development, implementation, and evaluation of a novel patient-oriented personalized preoperative risk communication eHealth application to empower patients, support shared decision making, and improve patient-centered outcomes. Development of this eHealth application will lead to an inclusively designed product tailored to the technology needs of elective surgery patients, who are typically older, and have limited technological expertise and comfort. The application will also be useful, in that it will communicate personalized risk estimates in a format consistent with best practices for risk communication to patients, and provide tools to engage shared discussions between patients and clinicians. Through implementation of the eHealth app, the Investigators will evaluate the effectiveness and value of personalized preoperative risk communication in improving knowledge, and satisfaction. The Investigators will also measure the acceptability of this process to patients and clinicians. Finally, the Investigators will test the feasibility of having a patient-oriented personalized risk communication application connect to the perioperative health system to identify high resource use patients prior to hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* English or French speaking
* Major elective, non-cardiac inpatient surgery

Exclusion Criteria:

* Unable to communicate in English or French
* Unable to consent without a Substitute Decision Maker
* Scheduled for non-elective surgery
* Patients having same-day surgery (outpatient surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit all consenting adults aged 18 or older seen in the Pre-Admission Unit prior to major elective, non-cardiac, inpatient surgery at The Ottawa Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hladkowicz E, Yachnin D, Boland L, Wilson K, McKinnon A, Hawrysh K, Hawrysh T, Bell C, Atkinson K, van Walraven C, Taljaard M, Thavorn K, Stacey D, Yang H, Pysyk C, Moloo H, Manuel D, MacDonald D, Lavallee LT, Gagne S, Forster AJ, Bryson GL, McIsaac DI. Evaluation of a preoperative personalized risk communication tool: a prospective before-and-after study. Can J Anaesth. 2020 Dec;67(12):1749-1760. doi: 10.1007/s12630-020-01809-y. Epub 2020 Sep 15. PMID 32929659

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Implementation Phase: Participants in this group (before the eHealth app is implemented in the Preadmission Unit (PAU)) will be English or French speaking patients, aged 18 and older, scheduled for major non-cardiac elective surgery.
  Patients will be recruited using standardized procedures, and process and outcome measures will be recorded using the same tools and methods in both study phases to decrease the risk of measurement and selection bias.
- Post-Implementation Phase: Participants in this group (after the eHealth app is implemented in the Preadmission Unit (PAU)) will be English or French speaking patients, aged 18 and older, scheduled for major non-cardiac elective surgery.
  Patient-oriented, personalized risk communication eHealth application: The application features simple and consistent design, large well-lit buttons that tolerate tremor, and simple language. The process will be applied in preoperative clinics at The Ottawa Hospital (TOH), where patients will be asked to provide their personal health history through a series of questions already used on our TOH preoperative health screener. These values will then populate the National Surgical Quality Improvement Program (NSQIP) Universal Risk Calculator, which we have calibrated to TOH data, to generate personalized risks of mortality, serious complications, and hospital length of stay. These risk estimates will be communicated directly to the patient using absolute risk estimates represented pictorially (best practice for risk communication to patients). Risk estimates will also be provided to the patient's clinician.
Period: Overall Study
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Started | 104 | 97
Completed | 90 | 93
Not Completed | 14 | 4
Not completed — Ineligible procedure, data error, patient declined because of timing, MD not consented | 14 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase | Total
Number analyzed (Participants) | 90 | 93 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14) | 64 (11) | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 34 | 82
  Male | 42 | 59 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] | 30 (8) | 30 (6) | 30 (7)

OUTCOME MEASURES:

1. Primary Outcome: Patient Knowledge
Description: Change in patient knowledge of their risk profile from before their Preadmission Unit (PAU). The questionnaire will not test perceived knowledge, but will test factual items specifically related to the patient's personalized risk profile.The pre- and post-appointment knowledge scores will be normalized on a 100 point scale [(questions correct/total questions)*100], scale scores will range from 0 to 100 (0=all questions incorrect, 100=all questions correct). A question was marked as correct if the patient's self-estimated risk and their model estimated risk were within the same range categoryHigher scores indicate higher levels of knowledge.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Number analyzed (Participants) | 90 | 93
score on a scale | 32.2 (28.5) | 53 (33.1)

2. Secondary Outcome: Anxiety
Description: Measured using the Short Form State-Trait Anxiety Inventory: at baseline and after the consultation using the short form State-Trait Anxiety Inventory, which is normalized to a 100-point scale. Scores can range from 20 to 80. Higher scores indicate greater levels of anxiety. Specifically, scores below 40 suggest minimal anxiety, while scores equal to or greater than 40 are considered clinically significant, indicating that the individual may be experiencing a heightened level of anxiety that could require further attention.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Number analyzed (Participants) | 90 | 93
score on a scale | 36.3 (11.6) | 29.4 (11.6)

3. Secondary Outcome: Patient Satisfaction- Likelihood to Recommend
Description: Patient experience will be assessed using a likelihood to recommend measurement based on a 10-point Likert scale (0 being not at all likely and 10 being extremely likely) to recommend the approach used to tell you about your surgical risk to a friend or family member) as recommended by the Institute for Healthcare Improvement's Triple Aim measurement guide.The value of the intervention will be defined using a patient-perceived equation as proposed by Morgan et al.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Number analyzed (Participants) | 90 | 93
score on a scale | 7.9 (2.5) | 8.9 (2.2)

4. Secondary Outcome: Patient Acceptability- Ease of Use
Description: Patient acceptability of the application will be assessed using a 5-point likert scale based on how easy it was to use (1 being the easiest and 5 being the hardest). The number of participants who find the application easy to use or very easy to use (gave a 1 or 2 on the likert scale) will be reported.
Time Frame: 1 day
Population: Participant feedback was not obtained for the pre-implementation phase as the app was not used.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Number analyzed (Participants) | 0 | 93
Participants | 0 | 87

5. Secondary Outcome: Clinician Change in Management
Description: Likelihood to change management will be measured using a 5-point scale, (1 strongly agree and 5 being strongly disagree) to change the management of the patient after reviewing the information provided by the personalized risk calculator. The number of participants that indicated that they strongly or moderately agreed (gave a score of 1 or 2 on the likert scale) that the application would lead to them making a change in anesthetic management will be reported.
Time Frame: 1 day
Population: The app was not used in the pre-implementation phase, therefore we did not obtain feedback from clinicians in the first phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Number analyzed (Participants) | 0 | 56
Participants | 0 | 2

6. Secondary Outcome: Clinician Acceptability
Description: Clinician acceptability of the application will be assessed using a 5-point likert scale (strongly disagree, moderately disagree, moderately agree, strongly agree or no opinion). The number of participants that strongly or moderately agreed that the personalized risk profiles were clear and unambiguous will be reported.
Time Frame: 1 day
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Number analyzed (Participants) | 0 | 56
Participants |  | 51

7. Secondary Outcome: Proportion of Patients for Whom a Risk Score Can be Calculated
Description: The proportion of patients for whom a risk score could be calculated - the number of participants who were able to have a risk score calculated out of the total sample will be reported (the number of participants who were able to provide the data required to calculate their personalized risk scores successfully using the application out of the total number of participants).
Time Frame: Through study completion for all participants, an average of one year
Population: The app was not used in the pre-implementation phase, therefore this is not applicable to the first phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Number analyzed (Participants) | 0 | 93
Participants | 0 | 93

8. Secondary Outcome: Proportion of Missing Data From the Patient-centered Health Questionnaire
Description: Proportion of missing data from the patient-centered health questionnaire - the number of participants with missing data for the patient-centered health questionnaire that is used to calculate risk out of the total sample will be reported.
Time Frame: Through study completion for all participants, an average of one year
Population: The app was not used in the pre-implementation phase, therefore this is not applicable to the first phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
Number analyzed (Participants) | 0 | 93
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Description: AEs were not expected or collected. The Total Number of Participants at Risk is 0 as serious and other [non-serious] adverse events were not collected or assessed as part of the study.
Arm/Group | Pre-Implementation Phase | Post-Implementation Phase
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We could not perform an individual patient randomized trial as the risk of contamination was deemed to be very high (we were concerned that exposure to a patient randomized to the PREDICT app would bias the clinician to access an online risk calculator [e.g., NSQIP online calculator] when caring for subsequent patients randomized to the control condition). As the knowledge assessed comes from the app, this could bias our results in favour of the PREDICT app.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT03422133/Prot_SAP_000.pdf